CLINICAL TRIAL: NCT04118400
Title: Ventilator Weaning Outcome Between Non-invasive Neural Adjusted Ventilator Assist and Nasal Continuous Positive Airway Pressure (or Intermittent Mandatory Ventilation) Modes in Premature Neonates
Brief Title: Ventilator Weaning Outcome Between NIV-NAVA and Nasal CPAP (or IMV ) Modes in Premature Neonates
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: N201907028
Record Dates: First submitted 2019-10-02; First posted 2019-10-08 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2019-10

CONDITIONS: Respiratory Distress Syndrome in Premature Infant

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental: NIN-NAVA: * Premature>30weeks with respiratory distress
  * PI to determine eligibility or exclusion
  * Randomize to either NIV-NAVA or Nasal CPAP (NIMV) 1:1 randomization
  * PI will not be blinded to the intervention (not feasible)
  * Place the catheter to optimize position
  * ABG or VBG to be obtained at 2 hrs. post NIV-NAVA
  * NIV-NAVA settings will be weaned or increased as the clinical situation demands and outlined in the protocol
  Interventions: Procedure: NIV-NAVA
- Active Comparator: Nasal CPAP or NIMV: * Premature>30weeks with respiratory distress
  * PI to determine eligibility or exclusion
  * Randomize to either NIV-NAVA or Nasal CPAP (NIMV) 1:1 randomization
  * PI will not be blinded to the intervention (not feasible)
  * Place the catheter to optimize position
  * ABG or VBG to be obtained at 2 hrs. post Nasal CPAP or NIMV
  * NCPAP or NIMV settings will be weaned or increased as the clinical situation demands and outlined in the protocol
  Interventions: Procedure: Nasal CPAP or NIMV mode

INTERVENTIONS:
Procedure: NIV-NAVA — NAVA mode during Non-invasive ventilation
  Groups: Experimental: NIN-NAVA
Procedure: Nasal CPAP or NIMV mode — Nasal CPAP or NIMV mode during Non-invasive ventilation
  Groups: Active Comparator: Nasal CPAP or NIMV

SUMMARY:
Premature neonates are prone to respiratory distress and need ventilator support because of the rapid breathing and large variations in respiratory patterns. The setting and adjustment of the ventilator for premature neonate is not easy, often resulting in poor patient-ventilator interaction, increased work of breathing, patient discomfort and delayed weaning . Recently, a new ventilation mode (NAVA; Neurally Adjusted Ventilatory Assist) mode, allows the respirator to provide a proportional ventilation mode based on the patients' diaphragm electrical activity, which was validated in many domestic and international clinical researches. The NAVA mode improves patient-ventilator interaction, reduces work of breathing and contributes to early weaning and extubation . When participating in this study, the neonate with receive a special oral tube placement, which is used to replace the original gastric tube to monitor the electrical activity of the diaphragm.

DETAILED DESCRIPTION:
Premature neonates are prone to respiratory distress and need ventilator support because of the rapid breathing and large variations in respiratory patterns. The setting and adjustment of the ventilator for premature neonate is not easy, often resulting in poor patient-ventilator interaction, increased work of breathing, patient discomfort and delayed weaning . Recently, a new ventilation mode (NAVA; Neurally Adjusted Ventilatory Assist) mode, allows the respirator to provide a proportional ventilation mode based on the patients' diaphragm electrical activity, which was validated in many domestic and international clinical researches. The NAVA mode improves patient-ventilator interaction, reduces work of breathing and contributes to early weaning and extubation . When participating in this study, the neonate with receive a special oral tube placement, which is used to replace the original gastric tube to monitor the electrical activity of the diaphragm. The aims of the study are: 1. To select the appropriate ventilation mode and parameters (for example, switch to NIV-NAVA mode); 2. To monitor intermittent apnea, bradycardia and the frequency of cyanosis, 3. To pay attention to the changes in maximum peak pressure, adjust appropriate pressure support, and avoid lung injury. The predicted outcomes of NAVA mode for premature neonate may include : 1. Measurement of the lower PIP value to maintain proper and synchronized ventilation; 2. Monitoring of the diaphragm activity (Edi) signal to evaluate the work of breathing and estimate the weaning time.

ELIGIBILITY:
Inclusion Criteria:

1. Premature >30week
2. Respiratory distress

Exclusion Criteria:

1. Premature < 30weeks
2. ENT contraindication: fistula
3. Contraindication with orogastric tube or nasogastric

Ages: 30 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature >30week and have Respiratory distress
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-10-31 (Actual); Primary Completion 2020-10-06 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Duration of mechanical ventilation | Until the date of discharge from ICU, up to 4 weeks
  Defined as the time from the start of mechanical ventilation, defined as either the time of in the ICU and until successful weaning mechanical ventilator, with successful weaning defined as ≥5 days of unassisted spontaneous breathing after .

SECONDARY OUTCOMES:
Daily patient physiological blood gas status | Until the date of discharge from ICU, up to 4 weeks
  Defined as daily PaO2/FiO2 from randomization until successful Weaning.
Length of ICU stay | Until the date of discharge from ICU, up to 4 weeks
  Defined as the duration of ICU admission from randomization to ICU discharge
Length of hospital stay | Until the date of discharge from ICU, up to 4 weeks
  Defined as the duration of hospital admission from randomization to hospital discharge
Difference in the number of patient ventilator asynchrony | Entire period of ventilatory support, an average of 7 days
  To assess the difference of number of patient ventilator asynchrony
Ventilation parameters: peak inspiratory pressure in NIV-NAVA | Entire period of ventilatory support, an average of 7 days
  Evolution of the following parameters: peak inspiratory pressure, tidal volume, PEEP, FiO2, Edi peak, Edi min )
Ventilation parameters : tidal volume in NIV-NAVA | through study completion, an average of 7 days
  Evolution of the following parameters: peak inspiratory pressure, tidal volume, PEEP, FiO2, Edi peak, Edi min )
Ventilation parameters : PEEP in NIV-NAVA | through study completion, an average of 7 days
  Evolution of the following parameters: peak inspiratory pressure, tidal volume, PEEP, FiO2, Edi peak, Edi min )
Ventilation parameters : FiO2 in NIV-NAVA | through study completion, an average of 7 days
  Evolution of the following parameters: peak inspiratory pressure, tidal volume, PEEP, FiO2, Edi peak, Edi min )
Ventilation parameters : Edi peak in NIV-NAVA | through study completion, an average of 7 days
  Evolution of the following parameters: peak inspiratory pressure, tidal volume, PEEP, FiO2, Edi peak, Edi min )
Ventilation parameters : Edi min in NIV-NAVA | through study completion, an average of 7 days
  Evolution of the following parameters: peak inspiratory pressure, tidal volume, PEEP, FiO2, Edi peak, Edi min )
Ventilation parameters : peak inspiratory pressure in NCPA (or NIMV) | through study completion, an average of 7 days
  Evolution of the following parameters: peak inspiratory pressure, tidal volume, PEEP, FiO2, PC Level, RR)
Ventilation parameters : tidal volume in NCPA(or NIMV) | through study completion, an average of 7 days
  Evolution of the following parameters: peak inspiratory pressure, tidal volume, PEEP, FiO2, PC, RR)
Ventilation parameters : PEEP in NCPA (or NIMV) | through study completion, an average of 7 days
  Evolution of the following parameters: peak inspiratory pressure, tidal volume, PEEP, FiO2, PCl, RR)
Ventilation parameters : FiO2 in NCPA or NIMV | through study completion, an average of 7 days
  Evolution of the following parameters: peak inspiratory pressure, tidal volume, PEEP, FiO2, PC, RR)
Ventilation parameters : pressure control level in NIMV | through study completion, an average of 7 days
  Evolution of the following parameters: peak inspiratory pressure, tidal volume, PEEP, FiO2, PC, RR)
Ventilation parameters : RR in NIMV | through study completion, an average of 7 days
  Evolution of the following parameters: peak inspiratory pressure, tidal volume, PEEP, FiO2, PC, RR)
Clinical parameters of Premature: heart rate in NIV-NAVA | through study completion, an average of 7days
  Evolution of clinical parameters (heart rate, respiratory rate, blood pressure) at the beginning and end of each period
Clinical parameters of Premature: respiratory rate in NIV-NAVA | through study completion, an average of 7days
  Evolution of clinical parameters (heart rate, respiratory rate, blood pressure) at the beginning and end of each period
Clinical parameters of Premature: SpO2 in NIV-NAVA | through study completion, an average of 7days
  Evolution of clinical parameters (SpO2) at the beginning and end of each period
Clinical parameters of Premature: blood pressure in NIV-NAVA | through study completion, an average of 7days
  Evolution of clinical parameters (heart rate, respiratory rate, blood pressure) at the beginning and end of each period
Clinical parameters of Premature: heart rate in NCPA(or NIMV) | through study completion, an average of 7days
  Evolution of clinical parameters (heart rate, respiratory rate, blood pressure) at the beginning and end of each period
Clinical parameters of Premature: respiratory rate in NCPA (or NIMV) | through study completion, an average of 7days
  Evolution of clinical parameters (heart rate, respiratory rate, blood pressure) at the beginning and end of each period
Clinical parameters of Premature: blood pressure in NCPA (or NIMV) | through study completion, an average of 7days
  Evolution of clinical parameters (heart rate, respiratory rate, blood pressure) at the beginning and end of each period
Clinical parameters of Premature: SpO2 in NCPAP(or NIMV) | through study completion, an average of 7days
  Evolution of clinical parameters (SpO2) at the beginning and end of each period

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-yu LI, Principal Investigator — Taipei Medical University Hospital, Taiwan, R.O.C
Locations (1):
- Hsin-yu LI, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting in January 2022
Access Criteria: starting in January 2022